CLINICAL TRIAL: NCT01214603
Title: A Phase 2 Study of LY2090314 in Participants With Acute Leukemia
Brief Title: A Study in Participants With Acute Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13370; I2H-MC-JWYB (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-09-29; First posted 2010-10-05 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-10

CONDITIONS: Leukemia
Keywords: Acute Myelogenous Leukemia, Acute Myeloid Leukemia, Acute; Leukemia, Leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — 3-(9-fluoro-2-(piperidin-1-ylcarbonyl)-1,2,3,4-tetrahydro(1,4)diazepino(6,7,1-hi)indol-7-yl)-4-imidazo(1,2-a)pyridin-3-yl-1H-pyrrole-2,5-dione

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2090314 (Experimental): Cohort 1: 40 milligrams (mg) LY2090314 administered on Days 1, 8, and 15 of a 28-day cycle for at least two (2) 28-day cycles. Participants experiencing clinical benefit may continue treatment until after the discontinuation criteria are met.
  Due to a protocol amendment on September 2010, the study added 2 additional treatment schedules/cohorts. Cohort 2: 40 mg dose given on Days 1, 5, and 9 of a 21-day cycle. Cohort 3: 40 mg dose given on Days 1, 5, 9, and 12 of a 21-day cycle. Participants experiencing clinical benefit may continue treatment until after the discontinuation criteria are met.
  Interventions: Drug: LY2090314

INTERVENTIONS:
Drug: LY2090314 — Administered intravenously

SUMMARY:
This study is a multicenter, non-randomized, open-label, Phase 2 study of intravenous LY2090314 in participants with acute leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have confirmed diagnosis of one of the following:

  * Acute myelogenous leukemia (AML) that is refractory or relapsed disease. If participants have acute promyelocytic leukemia (APL), they must have received prior all-trans retinoic acid and arsenic trioxide unless ineligible or intolerant to them
  * Untreated AML (de novo or arising from a myelodysplastic syndrome). In the opinion of the investigator, the participant should not be a candidate for standard therapy and a clinical trial is a preferred treatment option
* Have given written informed consent prior to any study-specific procedures
* Have adequate organ function including:

  * Hepatic: Bilirubin less than or equal to 1.5 times the upper limit of normal (ULN). Alkaline phosphatase (ALP) and transaminases [alanine aminotransferase (ALT) and aspartate aminotransferase (AST)] less than or equal to 5 times ULN
  * Renal: Serum creatinine less than or equal to the ULN. No known active renal disease. In rare cases, participants may enter treatment with a serum creatinine greater than the ULN as elevations of serum creatinine may be secondary to dehydration
* Have a performance status of less than or equal to 2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued all previous approved therapies for acute leukemia, including chemotherapy for at least 14 days, and recovered from the acute effects of therapy. Hydroxyurea used to control peripheral blast count is permitted within the first 2 cycles of treatment on study, but it must be stopped at least 24 hours before study drug administration in Cycle 3
* Are reliable and willing to be available for the duration of the study and are willing to follow study procedures
* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the trial and for 3 months following the last dose of study drug
* Females with childbearing potential must have had a negative urine or serum pregnancy test less than or equal to 7 days prior to the first dose of study drug
* Have an estimated life expectancy of greater than or equal to 6 weeks

Exclusion Criteria:

* Have received treatment within 14 days of the initial dose of study drug with an experimental agent for noncancer indications that has not received regulatory approval for any indication
* Participants with chronic myelogenous leukemia (CML) including blast crisis phase
* Participants with known central nervous system (CNS) leukemia by spinal fluid cytology or imaging
* Have serious pre-existing medical conditions (left to the discretion of the investigator)
* Have one of the following abnormalities: QTc (Fridericia corrected) interval >450 milliseconds (msec) on screening electrocardiogram (ECG), previous history of QTc prolongation with another medication that required discontinuation, congenital long QT syndrome, previous history of ventricular tachycardia or unexplained syncope, left bundle branch block, or chronic atrial fibrillation
* Have family history of long QT syndrome or sudden death due to ventricular arrhythmia
* Concomitant medication that may cause QTc prolongation or induce Torsades de Pointes at the time of study entry
* Have systolic blood pressure greater than or equal to 160 millimeter of mercury (mm Hg) and diastolic blood pressure greater than or equal to 100 mm Hg
* Have a serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease, as defined by the New York Heart Association Class II or higher or participants with a history of arrhythmia that is symptomatic or requires treatment
* Have uncorrected electrolyte disorders including potassium
* Have other active malignancy (with the exception of basal and squamous cell skin cancer) at time of study entry
* Have received an autologous or allogeneic stem-cell transplant within 75 days of the initial dose of study drug
* Have uncontrolled systemic infection
* Females who are pregnant or lactating
* Presence of clinical evidence of viral disease caused by human immunodeficiency virus, hepatitis B, or hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study had safety lead-in phase [40 milligrams (mg) LY2090314 administered using 3 treatment schedules]. Each cohort of participants had different schedule. Safety lead-in data determined if expansion phase opened to enrollment. No participant enrolled in expansion phase. Participants who completed 2 cycles of treatment considered study completers.
Groups:
- Cohort 1, 40 mg LY2090314: D1, D8, D15: LY2090314: 40 mg administered as an intravenous infusion over 60-minutes on Day (D)1, D8, and D15 for two 28-day cycles.
  If therapeutically beneficial, participants could continue additional treatment cycles until death, disease progression or other study discontinuation criteria were met.
- Cohort 2, 40 mg LY2090314: D1, D5, D9: LY2090314: 40 mg administered as an intravenous infusion over 60-minutes on D1, D5, and D9 for two 21-day cycles.
  If therapeutically beneficial, participants could continue additional treatment cycles until death, disease progression or other study discontinuation criteria were met.
- Cohort 3, 40 mg LY2090314: D1, D5, D9, D12: LY2090314: 40 mg administered as an intravenous infusion over 60-minutes on D1, D5, D9, and D12 for two 21-day cycles.
  If therapeutically beneficial, participants could continue additional treatment cycles until death, disease progression or other study discontinuation criteria were met.
Period: Overall Study
Arm/Group | Cohort 1, 40 mg LY2090314: D1, D8, D15 | Cohort 2, 40 mg LY2090314: D1, D5, D9 | Cohort 3, 40 mg LY2090314: D1, D5, D9, D12
Started | 7 | 6 | 7
Received at Least 1 Dose of LY2090314 | 7 | 6 | 7
Completed | 2 | 5 | 3
Not Completed | 5 | 1 | 4
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Progressive Disease | 4 | 1 | 3

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of LY2090314.
Groups:
- Cohort 1, 40 mg LY2090314: D1, D8, D15: LY2090314: 40 mg administered as an intravenous infusion over 60-minutes on D1, D8, and D15 for two 28-day cycles.
  If therapeutically beneficial, participants could continue additional treatment cycles until death, disease progression or other study discontinuation criteria were met.
- Total: Total of all reporting groups
Arm/Group | Cohort 1, 40 mg LY2090314: D1, D8, D15 | Cohort 2, 40 mg LY2090314: D1, D5, D9 | Cohort 3, 40 mg LY2090314: D1, D5, D9, D12 | Total
Number analyzed (Participants) | 7 | 6 | 7 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.3 (7.16) | 61.7 (14.98) | 67.6 (9.81) | 68.5 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5 | 10
  Male | 5 | 3 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 6 | 7 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 7 | 6 | 5 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 1 or More Study Drug-Related Adverse Events (AEs) or Any Serious AEs (SAEs)
Description: Drug-related events were defined as treatment-emergent serious and other non-serious AEs that were considered by the investigator to be related to study drug. A summary of serious and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through study completion [Cycle 9 plus 30 days post last dose (21-day or 28 day cycles)]
Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, 40 mg LY2090314: D1, D8, D15 | Cohort 2, 40 mg LY2090314: D1, D5, D9 | Cohort 3, 40 mg LY2090314: D1, D5, D9, D12
Number analyzed (Participants) | 7 | 6 | 7
Participants
  Study Drug-Related AE(s) | 6 | 5 | 6
  Study Drug-Related SAE(s) | 0 | 2 | 1

2. Secondary Outcome: Number of Participants With Best Response of Complete Response or Partial Response
Description: The Revised International Working Group criteria were used to determine the response for participants with acute myelogenous leukemia (AML). Complete response, also known as complete remission (CR) included the following categories: Morphologic CR defined as <5% blasts in an aspirate sample with marrow spicules and with a count of at least 200 nucleated cells, along with peripheral blood levels including platelets ≥100*10^9/Liter (L) and absolute neutrophil count (ANC) ≥1*10^9/L, Morphologic CR with incomplete blood count recovery (CRi), Cytogenetic CR, and Molecular CR. Partial response, also known as partial remission (PR) was defined as a decrease of at least 50% in blast count on the bone marrow aspirate. PR required all of the hematologic values for a CR but with a decrease of at least 50% in the percentage of blasts to 5% to 25% in the bone marrow aspirate.
Time Frame: Baseline to progressive disease (up to Cycle 9, 21-day or 28 day cycles)
Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, 40 mg LY2090314: D1, D8, D15 | Cohort 2, 40 mg LY2090314: D1, D5, D9 | Cohort 3, 40 mg LY2090314: D1, D5, D9, D12
Number analyzed (Participants) | 7 | 6 | 7
Participants
  CR | 0 | 0 | 0
  PR | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With Best Response of Complete Response or Partial Response
Description: The Revised International Working Group criteria were used to determine the response for participants with AML. Complete response, also known as complete remission (CR) included the following categories: Morphologic CR defined as <5% blasts in an aspirate sample with marrow spicules and with a count of at least 200 nucleated cells, along with peripheral blood levels including platelets ≥100*10^9/L and ANC ≥1*10^9/L, Morphologic CR with incomplete blood count recovery (CRi), Cytogenetic CR, and Molecular CR. Partial response, also known as partial remission (PR) was defined as a decrease of at least 50% in blast count on the bone marrow aspirate. PR required all of the hematologic values for a CR but with a decrease of at least 50% in the percentage of blasts to 5% to 25% in the bone marrow aspirate. Percentage of participants=[(number of participants with CR or PR)/(number of participants treated)]*100.
Time Frame: Baseline to progressive disease (up to Cycle 9, 21-day or 28 day cycles)
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, 40 mg LY2090314: D1, D8, D15 | Cohort 2, 40 mg LY2090314: D1, D5, D9 | Cohort 3, 40 mg LY2090314: D1, D5, D9, D12
Number analyzed (Participants) | 7 | 6 | 7
percentage of participants
  CR | 0.0 | 0.0 | 0.0
  PR | 0.0 | 0.0 | 0.0

4. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration-Time Curve From Time 0 to 8 Hours (h) Postdose [AUC(0-8)]
Description: AUC(0-8) was estimated from the plasma drug concentration time profile.
Time Frame: Cycle 1: D1 and/or D9 and/or D15 [predose, 30 minutes (during infusion), up to 24 h after infusion started (1 h, 2 h, 4 h, 6 h, 8 h, and 24 h)]
Population: Participants who received at least 1 dose of study drug and had sufficient postdose samples collected to allow estimation of the PK parameters using noncompartmental methods of analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Units Other Than Participants: Profiles
Groups:
- Entire Study Population: All participants who received at least 1 dose of LY2090314 regardless of the cohort to which they were enrolled.
  Cohort 1: LY2090314: 40 mg administered as an intravenous infusion over 60-minutes on D1, D8, and D15 for two 28-day cycles.
  Cohort 2: LY2090314: 40 mg administered as an intravenous infusion over 60-minutes on D1, D5, and D9 for two 21-day cycles.
  Cohort 3: LY2090314: 40 mg administered as an intravenous infusion over 60-minutes on D1, D5, D9, and D12 for two 21-day cycles.
  If therapeutically beneficial, participants could continue additional treatment cycles until death, disease progression or other study discontinuation criteria were met.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 13
Number analyzed (Profiles) | 14
nanograms*hours per milliliter (ng*h/mL) | 898 (47)

5. Secondary Outcome: PK: AUC From Time 0 to Infinity [AUC(0-inf)]
Description: AUC(0-inf) was estimated from the plasma drug concentration time profile.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Units Other Than Participants: Profiles
Arm/Group | Entire Study Population
Number analyzed (Participants) | 3
Number analyzed (Profiles) | 3
ng*h/mL | 963 (46.4)

6. Secondary Outcome: PK: Maximum Concentration (Cmax)
Description: Cmax is the maximum observed concentration estimated from the plasma drug concentration time profile.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Units Other Than Participants: Profiles
Arm/Group | Entire Study Population
Number analyzed (Participants) | 20
Number analyzed (Profiles) | 36
nanograms per milliliter (ng/mL) | 476 (56.5)

7. Secondary Outcome: Percent Change From Predose Beta (β)-Catenin Levels
Description: Percent change=[(β-catenin level postdose-predose level)/(predose β-catenin levels)]*100. Participants in Cohort 1 had β-catenin samples collected on Cycle 1: D1, D8, and D15, and Cycles 2 through 9: D1. Participants in Cohort 2 had β-catenin samples collected on Cycle 1: D1, D5, and D9 and Cycles 2 through 9: D1. Participants in Cohort 3 had β-catenin samples collected on Cycle 1: D1, D5, D9, and D12 and Cycles 2 through 9: D1.
Time Frame: Cycle 1: D1 and D9 (predose, 1 h, 2 h, 4 h, 8 h, and 24 h after infusion started); Cycle 1: D5, D8, and D12 and C2 through C9: D1 (predose, 2 h after infusion started); Cycle 1: D15 (predose, 1 h, 2 h, 4 h, and 8 h after infusion started)
Population: Participants who received at least 1 dose of study drug and had a predose and at least 1 postdose β-catenin sample collected.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Entire Study Population
Number analyzed (Participants) | 18
percent change
  Cycle 1, Day 1, 1 h postdose | 557.4 (397.49)
  Cycle 1, Day 1, 2 h postdose | 513.7 (284.19)
  Cycle 1, Day 1, 4 h postdose: number analyzed (Participants) | 17
  Cycle 1, Day 1, 4 h postdose | 547.6 (342.89)
  Cycle 1, Day 1, 8 h postdose: number analyzed (Participants) | 15
  Cycle 1, Day 1, 8 h postdose | 285.7 (421.91)
  Cycle 1, Day 1, 24 h postdose: number analyzed (Participants) | 11
  Cycle 1, Day 1, 24 h postdose | 83.6 (141.96)
  Cycle 1, Day 5, 2 h postdose: number analyzed (Participants) | 12
  Cycle 1, Day 5, 2 h postdose | 817.2 (576.25)
  Cycle 1, Day 8, 2 h postdose: number analyzed (Participants) | 7
  Cycle 1, Day 8, 2 h postdose | 343.2 (216.26)
  Cycle 1, Day 9, 1 h postdose: number analyzed (Participants) | 10
  Cycle 1, Day 9, 1 h postdose | 736.1 (831.56)
  Cycle 1, Day 9, 2 h postdose: number analyzed (Participants) | 10
  Cycle 1, Day 9, 2 h postdose | 746.5 (728.22)
  Cycle 1, Day 9, 4 h postdose: number analyzed (Participants) | 8
  Cycle 1, Day 9, 4 h postdose | 684.3 (630.99)
  Cycle 1, Day 9, 8 h postdose: number analyzed (Participants) | 6
  Cycle 1, Day 9, 8 h postdose | 141.2 (133.13)
  Cycle 1, Day 9, 24 h postdose: number analyzed (Participants) | 3
  Cycle 1, Day 9, 24 h postdose | 9.1 (99.14)
  Cycle 1, Day 12, 2 h postdose: number analyzed (Participants) | 6
  Cycle 1, Day 12, 2 h postdose | 837.8 (496.95)
  Cycle 1, Day 15, 1 h postdose: number analyzed (Participants) | 6
  Cycle 1, Day 15, 1 h postdose | 362.3 (246.81)
  Cycle 1, Day 15, 2 h postdose: number analyzed (Participants) | 6
  Cycle 1, Day 15, 2 h postdose | 470.6 (296.31)
  Cycle 1, Day 15, 4 h postdose: number analyzed (Participants) | 6
  Cycle 1, Day 15, 4 h postdose | 575.5 (422.33)
  Cycle 1, Day 15, 8 h postdose: number analyzed (Participants) | 5
  Cycle 1, Day 15, 8 h postdose | 474.2 (499.30)
  Cycle 2, Day 1, 2 h postdose: number analyzed (Participants) | 11
  Cycle 2, Day 1, 2 h postdose | 429.1 (339.86)
  Cycle 3, Day 1, 2 h postdose: number analyzed (Participants) | 5
  Cycle 3, Day 1, 2 h postdose | 348.5 (458.67)
  Cycle 4, Day 1, 2 h postdose: number analyzed (Participants) | 4
  Cycle 4, Day 1, 2 h postdose | 408.5 (291.78)
  Cycle 5, Day 1, 2 h postdose: number analyzed (Participants) | 4
  Cycle 5, Day 1, 2 h postdose | 186.3 (188.34)
  Cycle 6, Day 1, 2 h postdose: number analyzed (Participants) | 4
  Cycle 6, Day 1, 2 h postdose | 80.0 (77.57)
  Cycle 7, Day 1, 2 h postdose: number analyzed (Participants) | 3
  Cycle 7, Day 1, 2 h postdose | 151.3 (155.60)
  Cycle 8, Day 1, 2 h postdose: number analyzed (Participants) | 2
  Cycle 8, Day 1, 2 h postdose | 418.6 (357.18)
  Cycle 9, Day 1, 2 h postdose: number analyzed (Participants) | 1
  Cycle 9, Day 1, 2 h postdose | 83.1 (NA) — Only 1 participant included in the analysis, therefore standard deviation is not calculable.

8. Secondary Outcome: Number of Participants Who Died
Description: The number of participants who died while on study treatment and the number of participants who died during the 30-day follow-up (30 days post last dose) are reported.
Time Frame: Baseline through study completion [Cycle 9 plus 30 days post last dose (21-day or 28 day cycles)]
Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, 40 mg LY2090314: D1, D8, D15 | Cohort 2, 40 mg LY2090314: D1, D5, D9 | Cohort 3, 40 mg LY2090314: D1, D5, D9, D12
Number analyzed (Participants) | 7 | 6 | 7
Participants
  Death On Study, Prior To Cycle 2 Completion | 1 | 0 | 0
  Death On Study, Post Cycle 2 Completion | 0 | 1 | 0
  Death During 30-Day Follow-Up | 2 | 1 | 0

ADVERSE EVENTS:
Arm/Group | Cohort 1, 40 mg LY2090314: D1, D8, D15 | Cohort 2, 40 mg LY2090314: D1, D5, D9 | Cohort 3, 40 mg LY2090314: D1, D5, D9, D12
Serious Adverse Events (participants affected / at risk) | 4/7 | 5/6 | 6/7
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, 40 mg LY2090314: D1, D8, D15 (N=7) | Cohort 2, 40 mg LY2090314: D1, D5, D9 (N=6) | Cohort 3, 40 mg LY2090314: D1, D5, D9, D12 (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (3)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac ventricular disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ileitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1, 40 mg LY2090314: D1, D8, D15 (N=7) | Cohort 2, 40 mg LY2090314: D1, D5, D9 (N=6) | Cohort 3, 40 mg LY2090314: D1, D5, D9, D12 (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Halo vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal exudates (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 3 (4)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 2 (3) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nodule (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood fibrinogen decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 1 (1) | 2 (3)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 0/5 (0) | 1/3 (1) | 0/2 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
An interim data review was performed after 6 participants in the safety lead-in completed 1 cycle of therapy. Based on the interim safety results, the expansion cohort was not opened to enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days